CLINICAL TRIAL: NCT03850652
Title: Can Prebiotics Support the Treatment of Mild Iron Deficiency by Iron Supplementation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gemma Walton (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Sponsor-Investigator, Gemma Walton, Lecturer in Metagenomics; Principal Investigator, University of Reading
Organization: University of Reading (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: UREC 18/56
Record Dates: First submitted 2019-02-13; First posted 2019-02-22 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: Iron Supplementation; Prebiotics; Microbiota
MeSH Terms: interventions — Prebiotics; Iron-Dextran Complex; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic (Synergy-1) (Active Comparator): Prebiotic (Synergy-1) + Iron supplement
  Interventions: Dietary Supplement: Prebiotic (Synergy-1) + Iron supplement
- Maltodextrin (Placebo Comparator): Placebo (Maltodextrin) + Iron Supplement
  Interventions: Dietary Supplement: Placebo (Maltodextrin) + Iron Supplement

INTERVENTIONS:
Dietary Supplement: Prebiotic (Synergy-1) + Iron supplement — In addition, participants will be required to take one 7 g sachet of prebiotic food supplement daily. In addition, participants will be required to take one daily tablet of a generic, iron supplement (200 mg FeSO4 equivalent to 65 mg iron) (provided by pharmacy).
  Arms: Prebiotic (Synergy-1)
Dietary Supplement: Placebo (Maltodextrin) + Iron Supplement — participants will be required to take one 7 g sachet of placebo (maltodextrin) daily. In addition, participants will be required to take an iron supplement (200 mg FeSO4 equivalent to 65 mg iron) (provided by pharmacy).
  Arms: Maltodextrin

SUMMARY:
The first aim of this study is to investigate if daily administration of the prebiotic Synergy-1 (a commercial product consisting of oligofructose-enriched inulin) together with a common iron supplement (ferrous sulphate) during 4 weeks, in premenopausal non-anaemic women with low ferritin levels, would mitigate the adverse effects of iron on the gut microbiota. The estimated absorption rate of the ferrous salts is 10-15%, therefore the unabsorbed iron will reach the colon where it could stimulate growth of non-beneficial bacterial species in the intestinal environment. By contrast, prebiotics function by specifically supporting growth of the typically-beneficial microorganism such as bifidobacteria. Inulin-type fructans (ITF) are well recognised in this way. The hypothesis to be tested is that prebiotic consumption will lead to a beneficial shift in the microbiota helping against the dysbiosis associated with iron supplementation.

DETAILED DESCRIPTION:
This will be a crossover, placebo controlled, and randomised pilot study in 15 pre-menopausal female individuals with ferritin levels below 40 mcg/l but normal hemoglobin (Hb) and C reactive protein (CRP). The study will last 12 weeks and consist of two separated 4-week randomised intervention treatment periods with a prebiotic (Synergy-1) or placebo (Maltodextrin) in combination with an iron supplement (FeSO4) separated by a 4-week wash-out period. Volunteers will take daily doses of an iron supplement and a prebiotic (Synergy-1) or placebo (Maltodextrin) during the trial excepting in the washout period where the iron supplement and prebiotic/placebo treatments will be discontinued.

This trial will investigate the effects of an iron supplement treatment in combination with a prebiotic food supplement or placebo food supplement. Participants will be required to take one daily tablet of a generic, iron supplement (200 mg FeSO4 equivalent to 65 mg iron) (provided by pharmacy). In addition, participants will be required to take one of the products (prebiotic or placebo) daily at the same time each day. The prebiotic food supplement (supplied by the Beneo company) is a chicory inulin powder produced in Belgium. It has been used in scores of human intervention studies with no adverse effects. Participants will be required to take one 7 g sachet of prebiotic food supplement daily. This will be reconstituted with water and participants will be encouraged to take the sachet at the same time each day. The placebo control food supplement will be maltodextrin. Maltodextrin is a standard placebo product for use in human studies involving prebiotics and has been used safely at this dose, in many trials by ourselves for the last 20 years. The products will be provided as a powder (served in sachets) and identical in texture and appearance. The Beneo company will produce and provide barcoded sachets, blinded to the investigators and volunteers. After all volunteers have completed their study visits and all samples have been analysed by researchers, Beneo will provide information about barcoded sachets. Compliance to food supplement (prebiotic or placebo) will be assessed by recording intake in gastrointestinal (GI) diaries and participants will also be asked to return any unused sachets to the researchers at the end of the each 4-week intervention periods. For participants to be considered compliant and therefore included in the study, they will be required to take the food supplement or placebo at least 6 out of every 7 days of the trial for the week period and return completed questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-50 years
* Gender: Female
* Volunteers agree to sign an informal written consent form
* General good health
* Have ferritin levels below 40 mcg/l
* Normal or borderline-low hemoglobin levels (>11.5g/dL)

Exclusion Criteria:

* Use of antibiotics, prebiotics or probiotics (in food products or as supplements), laxatives, anti-spasmodic, anti-diarrhoea drugs, (e.g. Orlistat, Lactulose) in the last 4 weeks prior to, or during the study period.
* Use of any iron supplement in the last 6 months prior to the study period.
* If participants have received bowel preparation for investigative procedures in the 4 weeks prior to the study.
* Surgical resection of any part of the bowel.
* If participants are taking any medication whose effectiveness could be reduced by the iron administration (e.g. Levodopa, Levothyroxine).
* If participants have any chronic gut disorder/disease, such as inflammatory bowel syndrome (IBS), inflammatory bowel disease (IBD), etc. or other conditions that might affect the gut environment, e.g. coeliac disease.
* If participants are taking any medication that could affect the iron absorption (e.g. lansoprazole, omeprazole).
* If participants are pregnant or are lactating.
* If participants have a body mass index (BMI) > 30 kg/m2.
* Severe allergy or any history of severe abnormal drug reaction, drug or alcohol abuse.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03-06 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the faecal microbiota composition by Next Generation Sequencing (NGS) | 12 weeks intervention
  Changes in composition of faecal microbiota attributable to prebiotic and iron intervention assessed by Next Generation Sequencing.
Changes in the concentration (mcg/g) of faecal calprotectin (gut inflammatory marker) during iron intervention using enzyme-linked immunosorbent assays (ELISAs). | 12 weeks intervention
  Gut inflammation will be evaluated measuring concentration (mcg/g) of calprotectin. Elevated faecal calprotectin indicates the migration of neutrophils to the intestinal mucosa, which occurs during intestinal inflammation
Changes in the concentration (pg/mL) of inflammatory markers in plasma during iron intervention using enzyme-linked immunosorbent assays (ELISAs). | 12 weeks intervention
  Gut inflammation will be also assessed measuring concentration (pg/mL) of gut inflammatory markers as plasma intestinal fatty acid-binding protein and cytokines from plasma (i.e interleukin 6, interleukin 10, tumor necrosis factor alpha). Samples will be analysed using enzyme-linked immunosorbent assays (ELISAs).
Changes in faecal microbiota activity measured by using Nuclear magnetic resonance spectroscopy (NMR) | 12 weeks intervention
  Changes in the metabolic profile during the intervention will be measured in urine and faecal samples by NMR.
Changes in faecal water genotoxicity of the volunteers during the intervention by comet assay (single cell gel electrophoresis assay using HT29 cells with Komet 5.5 software) | 12 weeks intervention
  Genotoxicity of volunteer faecal water will be measured at baseline and during intervention to determine whether prebiotic intervention can ameliorate iron-induced enterocyte genotoxicity. HT29 cells will be exposed to faecal waters, then single stranded breaks to the DNA will be quantified using Komet 5.5 software.

SECONDARY OUTCOMES:
Daily assessment of stool consistency | 12 weeks intervention
  Volunteers will keep a daily diary noting the consistency of the stools using the Bristol stool chart.
Daily assessment of gastrointestinal symptoms | 12 weeks intervention
  Volunteers will keep a daily diary recording abnormal pain, bloating or flatulence

CONTACTS AND LOCATIONS:
Overall Officials: Simon C Andrews, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data of faecal bacterial DNA may be made available to The European Bioinformatics Institute. This will help support other research in the field